CLINICAL TRIAL: NCT02579850
Title: 52-week, Double Blind, Randomized, 2 Active Parallel Arms Study of Fixed Combination CHF 5993 Administered vs Ultibro® in COPD Patients
Brief Title: 2-arm Parallel Group Study of Fixed Combination of CHF 5993 vs Ultibro® in COPD Patients
Acronym: TRIBUTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-05993AA1-08; 2014-001704-22 (EudraCT Number)
Record Dates: First submitted 2015-05-12; First posted 2015-10-20 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; COPD Exacerbation; EXACT-PRO
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF 5993 + Ultibro matched placebo (Experimental): Fixed triple therapy with BDP/FF/GB 100/6/12.5 mcg (CHF 5993) administered 2 puffs twice daily via pMDI + Fixed combination of indacaterol and of glycopyrronium (Ultibro® Breezhaler®) matched placebo administered once daily via DPI for 52-week treatment.
  Patient used to take pMDI medication using a spacer will be provided with a new spacer for the study.
  7 study visits including : central spirometry tests, Local laboratory, COPD assessment test (visit 1 only), Local laboratory Assessments Saint George's Respiratory Questionnaire EXACT-pro questionnaire
  Interventions: Drug: CHF 5993 + Ultibro matched placebo; Procedure: Central spirometry; Other: COPD assessment test; Procedure: Local laboratory Assessments; Other: Saint George's Respiratory Questionnaire; Other: EXACT-pro questionnaire
- Ultibro + CHF 5993 matched placebo (Active Comparator): Fixed combination of indacaterol 85 mcg and of glycopyrronium 43 mcg (Ultibro® Breezhaler®) administered once daily via DPI + Fixed triple therapy with BDP/FF/GB (CHF 5993) matched placebo administered 2 puffs twice daily via pMDI for 52-week treatment.
  Patient used to take pMDI medication using a spacer will be provided with a new spacer for the study.
  7 study visits including : central spirometry tests, Local laboratory, COPD assessment test (visit 1 only), Local laboratory Assessments, Saint George's Respiratory Questionnaire, EXACT-pro questionnaire
  Interventions: Drug: Ultibro + CHF 5993 matched placebo; Procedure: Central spirometry; Other: COPD assessment test; Procedure: Local laboratory Assessments; Other: Saint George's Respiratory Questionnaire; Other: EXACT-pro questionnaire

INTERVENTIONS:
Drug: CHF 5993 + Ultibro matched placebo — Active medication treatment CHF 5993 and Ultibro matched placebo administered twice a day
  Other Names: CHF 5993
  Arms: CHF 5993 + Ultibro matched placebo
Drug: Ultibro + CHF 5993 matched placebo — Active medication treatment Ultibro and CHF 5993 matched placebo administered twice a day
  Other Names: Ultibro Breezhaler
  Arms: Ultibro + CHF 5993 matched placebo
Procedure: Central spirometry — Central spirometry to assess forced expiratory volume at one second and forced vital capacity
Other: COPD assessment test — COPD assessment test (CAT) at visit 1
Procedure: Local laboratory Assessments — ECG + Standard Haematology and Biochemistry
Other: Saint George's Respiratory Questionnaire — Saint George's Respiratory Questionnaire
Other: EXACT-pro questionnaire — daily from randomization (Visit 2) to end of study (Visit 7)

SUMMARY:
The aim of the present study is to evaluate the superiority of the fixed triple therapy with BDP/FF/GB at a daily dose of 400/24/50 mcg respectively with that of Ultibro® Breezhaler® (DPI), fixed combination of indacaterol 85 mcg and of glycopyrronium 43 mcg in COPD patients.

DETAILED DESCRIPTION:
Outpatients attending the hospital clinics/study centres will be recruited. Patients with severe and very severe COPD airflow obstruction according to GOLD 2014 criteria. A total of approximately 2192 patients will need to be screened in order to obtain 1534 (767 per arm) randomized and evaluable patients. Approximately 200 sites will be involved worldwide.

Each patient will perform a total of 8 clinic visits (V0 to V7) during the study.

The Primary objective is to demonstrate the superiority of CHF 5993 pMDI over Ultibro® in terms of moderate and severe COPD exacerbation rate over 52 weeks of treatment.

The Secondary objectives are:

1. To evaluate the effect of CHF 5993 pMDI on other lung function parameters, patient's health status and clinical outcome measures;
2. To assess the safety and the tolerability of the study treatments.

A 2-week open-label run-in period under Ultibro® followed by a 52-week randomised treatment period.

The trial design will be optimised to measure exacerbation rates by using the Exacerbations of Chronic Pulmonary Disease Tool (EXACT), developed means of collecting patient-reported outcome (PRO) data, which helps to capture the frequency of exacerbations.

ELIGIBILITY:
Inclusion :

1. Male and female ≥ 40 years
2. Severe or very severe COPD diagnosed for at least 12 months
3. Current smokers or ex-smokers who quit smoking at least 6 months prior to screening visit, with a smoking history of at least 10 pack years
4. Post-bronchodilator FEV1 < 50% of the predicted normal value and a post-bronchodilator FEV1/FVC ratio < 0.7
5. Documented history of at least one exacerbation in the 12 months
6. Patient under double therapy for at least 2 months prior to screening. Double therapy will be defined by treatment with any of the following:

   Orally inhaled corticosteroid (ICS) and (long-acting beta2-agonist) LABA ICS and long-acting muscarinic antagonist (LAMA) Orally LABA and LAMA Monotherapy with LAMA for at least 2 months prior to screening
7. Symptomatic patient at screening with a CAT score ≥ 10.
8. Cooperative attitude and ability to use correctly the inhalers, the spacer AeroChamber Plus (only to patients who are using a spacer), the electronic devices with COPD questionnaire.

Exclusion :

1. Pregnant or lactating women and all women physiologically capable of becoming pregnant UNLESS are willing to use one or more of the reliable methods of contraception
2. Patient with a current clinical diagnosis of asthma with a physician-judged need for inhaled or oral corticosteroid therapy
3. Patient requiring use of the following medications:

   Course of systemic steroids > 3 days for COPD exacerbation in the 4 weeks prior to screening Course of antibiotics for COPD exacerbation > 7 days in the 4 weeks prior to screening Phosphodiesterase-4 inhibitor in the 4 weeks prior to screening Use of antibiotics for a lower respiratory tract infection in the 4 weeks prior to screening
4. COPD exacerbation requiring prescription of systemic corticosteroids and/or antibiotics or hospitalization during the run-in period
5. Patient treated with non-cardioselective β-blockers in the month preceding the screening or during the run-in period.
6. Patient treated with long-acting antihistamines unless taken at stable regimen at least 2 months prior to screening and to be maintained constant during the study or if taken as needed
7. Patient requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia
8. Known respiratory disorders other than COPD which may impact the efficacy of the study drug
9. Patient who have clinically significant cardiovascular condition
10. Patient with atrial fibrillation (AF): Paroxysmal atrial fibrillation, Persistent, Long standing or Permanent
11. Abnormal and clinically significant 12-lead ECG that results in active medical problem which may impact the safety of the patient
12. Patient whose ECG shows QTcF >450 ms for males or QTcF >470 ms for females at screening visit are not eligible (not applicable for patient with pacemaker)
13. Medical diagnosis of narrow-angle glaucoma, clinically relevant prostatic hypertrophy or bladder neck obstruction would prevent use of anticholinergic agents
14. History of hypersensitivity to M3 Antagonists, β2-agonist, corticosteroids or any of the excipients contained in any of the formulations used in the trial which may raise contra-indications or impact the efficacy of the study drug
15. Clinically significant laboratory abnormalities indicating a significant or unstable concomitant disease which may impact the efficacy or the safety of the study drug
16. Patients with hypokalaemia (serum potassium <3.5 mEq/L or 3.5 mmol/L) or uncontrolled hyperkalaemia
17. Unstable concurrent disease which may impact the results of the study
18. Patients with any history of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next six months (after V1) or with malignancy for which they are currently undergoing radiation therapy or chemotherapy
19. History of alcohol abuse or substance/drug abuse within 12 months prior to screening visit
20. Participation in another clinical trial if investigational drug was received less than 8 weeks prior to screening visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1532 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Moderate and severe COPD exacerbation rate over 52 weeks of treatment | 1 year
  Exacerbations will be evaluated at each study visit and collected using EXACT-PRO filled-in by patient every day throughout the study

SECONDARY OUTCOMES:
Time to first moderate to severe COPD exacerbation | 1 year
Rate of severe COPD exacerbation over 52 weeks of treatment | 1 year
Rate of moderate COPD exacerbation over 52 weeks of treatment | 1 year
Change from Baseline at each visit and over the entire treatment period in pre-dose morning FEV1 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mario Scuri, MD, Study Chair — Chiesi Farmaceutici S.p.A.; Nicolas Roche, Pr, Principal Investigator — Hopitaux Universitaires Paris Centre - Groupe Hospitalier Cochin
Locations (1):
- Chiesi Farmaceutici S.p.A., Parma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- [Background] Vanfleteren L, Fabbri LM, Papi A, Petruzzelli S, Celli B. Triple therapy (ICS/LABA/LAMA) in COPD: time for a reappraisal. Int J Chron Obstruct Pulmon Dis. 2018 Dec 12;13:3971-3981. doi: 10.2147/COPD.S185975. eCollection 2018. PMID 30587953
- [Background] Singh D, Fabbri LM, Vezzoli S, Petruzzelli S, Papi A. Extrafine triple therapy delays COPD clinically important deterioration vs ICS/LABA, LAMA, or LABA/LAMA. Int J Chron Obstruct Pulmon Dis. 2019 Feb 28;14:531-546. doi: 10.2147/COPD.S196383. eCollection 2019. PMID 30880943
- [Background] Singh D, Fabbri LM, Corradi M, Georges G, Guasconi A, Vezzoli S, Petruzzelli S, Papi A. Extrafine triple therapy in patients with symptomatic COPD and history of one moderate exacerbation. Eur Respir J. 2019 May 18;53(5):1900235. doi: 10.1183/13993003.00235-2019. Print 2019 May. PMID 30792343
- [Background] Papi A, Petruzzelli S, Vezzoli S, Georges G, Fabbri LM. Triple therapy for all patients with severe symptomatic COPD at risk of exacerbations. Eur Respir J. 2019 Apr 18;53(4):1900147. doi: 10.1183/13993003.00147-2019. Print 2019 Apr. No abstract available. PMID 31000665
- [Result] Papi A, Vestbo J, Fabbri L, Corradi M, Prunier H, Cohuet G, Guasconi A, Montagna I, Vezzoli S, Petruzzelli S, Scuri M, Roche N, Singh D. Extrafine inhaled triple therapy versus dual bronchodilator therapy in chronic obstructive pulmonary disease (TRIBUTE): a double-blind, parallel group, randomised controlled trial. Lancet. 2018 Mar 17;391(10125):1076-1084. doi: 10.1016/S0140-6736(18)30206-X. Epub 2018 Feb 9. PMID 29429593
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2014-001704-22/results
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/33_CSR_Synopsis_CCD-05993AA1-08.pdf